CLINICAL TRIAL: NCT04744935
Title: Optical Coherence Tomography Guided Laser Treatment of Basal Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Zachary (Other)
Responsible Party: Sponsor-Investigator, Christopher Zachary, Professor and Chair of the UCI Department of Dermatology, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20205664
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Basal Cell Carcinoma; Superficial Basal Cell Carcinoma; Nodular Basal Cell Carcinoma
Keywords: Basal cell carcinoma; Superficial basal cell carcinoma; Nodular basal cell carcinoma; Optical coherence tomography; OCT; Laser
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard (Active Comparator): 1064 Long-pulse Nd:YAG laser Fluence: 120 J/cm2 Number of passes: Single Spot size: 2 cm Pulse width: 8-10 msec
  Interventions: Device: 1064 nm long-pulse Nd:YAG laser
- Slow (Active Comparator): 1064 Long-pulse Nd:YAG laser Fluence: 20-30 J/cm2 Number of passes: Multiple Spot size: 2 cm Pulse width: 8-10 msec
  Interventions: Device: 1064 nm long-pulse Nd:YAG laser

INTERVENTIONS:
Device: 1064 nm long-pulse Nd:YAG laser — BCC lesion will be treated with long-pulse 1064 laser, with surface temperature monitored by infrared camera.

SUMMARY:
Optical coherence tomography guided laser treatment of basal cell carcinoma

DETAILED DESCRIPTION:
The purpose of this pilot study is to examine the treatment basal cell carcinoma (BCC) with laser technology under the guidance of optical coherence tomography imaging (OCT). The laser modality that we plan to use is the long-pulse Nd:YAG 1064nm laser, which is a non-ablative laser already shown to effectively treat BCC. Laser treatment of BCC has limited precedent in the literature, but the addition of OCT has the opportunity to enhance outcomes by better targeting the treatment and permitting more precise monitoring of clearance. We propose to use OCT imaging to guide the laser treatment to achieve optimal efficacy with minimized side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and carry out subject instructions or be represented by a legally authorized guardian or representative
* Ages 18 and older
* Seeks and is scheduled for treatment of a BCC previously confirmed with biopsy

Exclusion Criteria:

Any of the following will exclude participation in the study:

* Inability to understand and/or carry out instructions
* Patients with a BCC lesion that requires excision. This would include relatively large lesions (>2.5 cm diameter), lesions that penetrate deep into the skin beyond the depth of the OCT image capture, high risk lesions as defined by the American Academy of Dermatology as recurrent and sclerosing subtype BCC, or metastases.
* Patients with periocular BCCs which might expose the patient to risk of damage to eyes from the laser.
* BCCs on legs due to their tendency towards poor wound healing.
* Pregnancy
* Patients unable to follow-up for the full 12 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete clearance of BCC lesion | 1 year
  Those whose lesion is not in a cosmetically sensitive area will undergo a skin biopsy for histological confirmation of OCT results.

SECONDARY OUTCOMES:
Cosmetic outcome | 1 year
  We assess cosmetic outcome and any adverse effects of the laser treatment as a result of the laser treatment, rated on a 0-4 Likert scaleworst cosmetic outcome and 4 resembling normal skin, upon follow-up of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Zachary, MBBS FRCP, Principal Investigator — University of California, Irvine
Locations (1):
- UCI Health Gottschalk Medical Plaza, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No